CLINICAL TRIAL: NCT04365257
Title: Alpha-1 Adrenergic Receptor Antagonism to Prevent COVID-19 Cytokine Storm Syndrome and Acute Respiratory Distress Syndrome: A Randomized Study Comparing the Efficacy of Prazosin vs. Standard of Care for SARS-CoV-2 Infection
Brief Title: Prazosin to Prevent COVID-19 (PREVENT-COVID Trial)
Acronym: PREVENT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: Johns Hopkins University (Other)
Collaborators: Fast Grants (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00246659; COV2001 (Other: Johns Hopkins University)
Record Dates: First submitted 2020-04-24; First posted 2020-04-28 (Actual); Results first posted 2023-01-31 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-03

CONDITIONS: COVID-19
Keywords: SARS-CoV-2; Coronavirus disease 2019; COVID-19; Cytokine Storm Syndrome; Acute Respiratory Distress Syndrome; Prazosin; Alpha-1 receptor antagonist
MeSH Terms: conditions — COVID-19; Cytokine Release Syndrome; Respiratory Distress Syndrome | interventions — Prazosin; Adrenergic alpha-1 Receptor Antagonists; Adrenergic alpha-Antagonists; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Prazosin (Experimental): 1. Prazosin 1mg given to observe if medication is tolerated or if signs or symptoms of hypotension develop (e.g. dizziness, lightheadedness).
  2. If the patient remains asymptomatic and BP >110/60 mmHg, prazosin is continued at 1mg every 8 hours (q8h).
  3. Day 3: If the patient remains asymptomatic and BP >110/60 mmHg, increase dose to 2mg q8h.
  4. Day 6: If the patient remains asymptomatic and BP >110/60 mmHg, increase dose to 5mg q8h.
  5. If the BP is <100/60 mmHg at any time, the next dose should be held, and patient continues with the highest previously tolerated dose 8 hours later.
  6. If the patient did not tolerate dose escalation to 5mg q8h, one attempt is made to increase dose to 3mg q8h. If this is not tolerated, the patient continues with the highest previously tolerated dose 8 hours later.
  If BP monitoring is not available, repeated occurrences of postural dizziness should trigger drug dose reduction or BP monitoring.
  Interventions: Drug: Prazosin
- Standard of care (Active Comparator): Subjects randomized to this arm will receive standard of care.
  Interventions: Other: Standard of care

INTERVENTIONS:
Drug: Prazosin — Participants in this arm will receive the study drug as outlined in the arm description.
  Other Names: Minipress; alpha-1 adrenergic receptor antagonist; alpha blocker
  Arms: Prazosin
Other: Standard of care — Participants in this arm will receive standard of care.
  Arms: Standard of care

SUMMARY:
The purpose of this study is to assess the efficacy and safety of prazosin to prevent cytokine storm syndrome and severe complications in hospitalized patients with Coronavirus disease 2019 (COVID-19).

DETAILED DESCRIPTION:
In Coronavirus disease 2019 (COVID-19), severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) elicits an exuberant local or systemic immune response ('hyperinflammation') in the lung and other sites of viral replication, compromising organ function and leading to high morbidity and mortality. Emerging evidence suggests that a subset of patients with COVID-19 develops a cytokine storm syndrome that is associated with elevation of pro-inflammatory cytokines.

Catecholamines enhance inflammatory injury by augmenting the production of IL-6 and other cytokines through a self-amplifying feed-forward loop in immune cells that requires alpha-1 adrenergic receptor (⍺1-AR) signaling. The ⍺1-AR antagonist prazosin prevents cytokine storm and markedly increased survival following inflammatory stimuli in preclinical models. In a retrospective study of outcomes in acute respiratory distress syndrome or pneumonia, patients who were taking ⍺1-AR antagonists had significantly lower probability of needing invasive mechanical ventilation and dying in the hospital compared to non-users.

Prazosin may blunt surges in catecholamines and self-amplifying cytokine production (including interleukin 6) and, as an early preemptive therapy in patients prior to disease progression, may prevent cytokine storm syndrome and severe complications of COVID-19.

In this study, patients with positive SARS-CoV-2 testing who are hospitalized (but are not requiring more than 4 liters/minute of supplemental oxygen by nasal cannula) will be screened for eligibility. Patients who provide informed consent and meet eligibility requirements will be randomized in a 1:1 ratio to receive either prazosin or standard of care. Participants randomized to the study drug will receive prazosin for 28 days and all patients will be followed for a total of 60 days to capture outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 45 years of age or older
* Provision of informed consent
* Subjects who tested positive for SARS-CoV-2 AND have clinical symptoms of COVID-19* AND have been hospitalized, but are not requiring more than 4 liters/minute of supplemental oxygen by nasal cannula and are not requiring ICU/CCU-level care at time of enrollment

(*)Acute respiratory tract infection (sudden onset of at least one of the following: fever, chills, sore throat, myalgia, diarrhea, cough, or shortness of breath) AND with no other etiology that fully explains the clinical presentation

Exclusion Criteria:

* Female subjects who identify as pregnant, self-reported positive pregnancy testing, or who are breastfeeding during the study period
* Age >85 years
* Known history of known orthostatic hypotension, unexplained history of syncope, postural orthostatic tachycardia syndrome (POTS), neurally-mediated hypotension, heart failure, myocardial infarction, stable or unstable angina, history of coronary artery bypass surgery, stroke, carotid artery disease, or moderate to severe mitral or aortic stenosis
* Current use of tocilizumab, sarilumab, siltuximab, lopinavir/ritonavir, remdesivir, favipiravir, alpha-blockers, combined alpha/beta blockers (carvedilol, labetalol), sotalol, clonidine, phosphodiesterase type 5 inhibitors, asenapine, or alpha-methyldopa
* Need for vasopressors, inotropes, or intra-aortic balloon pump at time of enrollment
* Allergy or intolerance to quinazolines (including prazosin)
* Requires oxygen supplementation beyond 4 liters of oxygen/minute per nasal cannula at time of enrollment (i.e. not requiring oxygenation by non-rebreather, high-flow nasal cannula, CPAP/BiPAP, or invasive mechanical ventilation)
* Patients who are in the custody of state or federal entities (prisoners)

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-05-13 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chetan Bettegowda, MD/PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Prazosin: 1. Prazosin 1mg given to observe if medication is tolerated or if signs or symptoms of hypotension develop (e.g. dizziness, lightheadedness).
  2. If the patient remains asymptomatic and BP >110/60 mmHg, prazosin is continued at 1mg every 8 hours (q8h).
  3. Day 3: If the patient remains asymptomatic and BP >110/60 mmHg, increase dose to 2mg q8h.
  4. Day 6: If the patient remains asymptomatic and BP >110/60 mmHg, increase dose to 5mg q8h.
  5. If the BP is <100/60 mmHg at any time, the next dose should be held, and patient continues with the highest previously tolerated dose 8 hours later.
  6. If the patient did not tolerate dose escalation to 5mg q8h, one attempt is made to increase dose to 3mg q8h. If this is not tolerated, the patient continues with the highest previously tolerated dose 8 hours later.
  If BP monitoring is not available, repeated occurrences of postural dizziness should trigger drug dose reduction or BP monitoring.
  Prazosin: Participants in this arm will receive the study drug as outlined in the arm description.
Period: Overall Study
Arm/Group | Prazosin | Standard of Care
Started | 3 | 2
Completed | 1 | 1
Not Completed | 2 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Patient Noncompliance | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prazosin | Standard of Care | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 0 | 3
  >=65 years | 0 | 2 | 2
Age, Continuous [Median (Full Range); unit: years] | 53.3 [47 to 57] | 71 [71 to 71] | 60.4 [47 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Death
Description: Number of participants in each arm who expire.
Time Frame: up to day 60
Measure: Count of Participants; unit: Participants
Arm/Group | Prazosin | Standard of Care
Number analyzed (Participants) | 3 | 2
Participants | 0 | 0

2. Primary Outcome: Hospitalized, Requiring Mechanical Ventilation and/or High Flow Nasal Cannula and/or ICU/CCU Admission (or Equivalent) and/or ECMO
Description: Number of participants in each arm who are hospitalized and requiring mechanical ventilation and/or high flow nasal cannula and/or ICU/CCU admission (or equivalent) and/or ECMO.
Time Frame: up to day 60
Measure: Count of Participants; unit: Participants
Arm/Group | Prazosin | Standard of Care
Number analyzed (Participants) | 3 | 2
Participants | 0 | 1

3. Primary Outcome: Hospitalized, Requiring Supplemental Oxygen, Not Requiring ICU/CCU Level Care (or Interventions Listed Under Outcome 2)
Description: Number of participants in each arm who are hospitalized and requiring supplemental oxygen, not requiring ICU/CCU level care (or interventions listed under Outcome 2).
Time Frame: up to day 60
Measure: Count of Participants; unit: Participants
Arm/Group | Prazosin | Standard of Care
Number analyzed (Participants) | 3 | 2
Participants | 2 | 1

4. Primary Outcome: Cumulative Incidence of Grade 3 and 4 Adverse Events
Description: Number of participants in each arm who develop grade 3 and 4 adverse events during the study period.
Time Frame: up to day 60
Measure: Count of Participants; unit: Participants
Arm/Group | Prazosin | Standard of Care
Number analyzed (Participants) | 3 | 2
Participants | 0 | 0

5. Primary Outcome: Number of Participants With Serious Adverse Events
Description: Number of participants in each arm who develop serious adverse events during the study period.
Time Frame: up to day 60
Measure: Count of Participants; unit: Participants
Arm/Group | Prazosin | Standard of Care
Number analyzed (Participants) | 3 | 2
Participants | 0 | 0

6. Primary Outcome: Incidence of Symptomatic Hypotension or Hypotension Requiring Cessation of Prazosin
Description: Number of participants in each arm who develop symptomatic hypotension (systolic blood pressure <90 mmHg) or hypotension requiring cessation of prazosin.
Time Frame: up to day 60
Measure: Count of Participants; unit: Participants
Arm/Group | Prazosin | Standard of Care
Number analyzed (Participants) | 3 | 2
Participants | 0 | 0

7. Secondary Outcome: Number of Participants With Laboratory Abnormalities in Peripheral Blood
Description: Number of participants with laboratory abnormalities in peripheral blood (Lymphopenia, leukocytosis, anemia, thrombocytopenia, creatinine, AST/ALT, troponin I, pro-BNP, D-dimer, ferritin, interleukin (IL-6), soluble IL-2 receptor.
Time Frame: up to day 60
Measure: Count of Participants; unit: Participants
Arm/Group | Prazosin | Standard of Care
Number analyzed (Participants) | 3 | 2
Participants | 0 | 0

8. Secondary Outcome: Duration of Laboratory Abnormalities in Peripheral Blood
Description: Number of days with laboratory abnormalities in peripheral blood (Lymphopenia, leukocytosis, anemia, thrombocytopenia, creatinine, AST/ALT, troponin I, pro-BNP, D-dimer, ferritin, interleukin (IL-6), soluble IL-2 receptor.
Time Frame: up to day 60
Population: Data was not collected because no participant had laboratory abnormalities in peripheral blood.
Arm/Group | Prazosin | Standard of Care
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Number of Participants With Laboratory Abnormalities in Plasma
Description: Number of participants with laboratory abnormalities in fractionated plasma catecholamines and plasma metanephrines.
Time Frame: up to day 60
Measure: Count of Participants; unit: Participants
Arm/Group | Prazosin | Standard of Care
Number analyzed (Participants) | 3 | 2
Participants | 0 | 0

10. Secondary Outcome: Duration of Laboratory Abnormalities in Plasma
Description: Number of days with laboratory abnormalities in fractionated plasma catecholamines and plasma metanephrines.
Time Frame: up to day 60
Population: Data was not collected because no participant had laboratory abnormalities in plasma.
Arm/Group | Prazosin | Standard of Care
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 60 days
Arm/Group | Prazosin | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 1/3 | 1/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prazosin (N=3) | Standard of Care (N=2)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
dizziness (General disorders) | 0 (0) | 1 (1)
urinary urgency (Renal and urinary disorders) | 0 (0) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1) | 0 (0)
Hypoxia during the night (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-12): https://cdn.clinicaltrials.gov/large-docs/57/NCT04365257/Prot_SAP_000.pdf